CLINICAL TRIAL: NCT04747470
Title: A Phase 1b Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of GS-3583, a FLT3 Agonist Fc Fusion Protein, in Subjects With Advanced Solid Tumors
Brief Title: Study to Assess the Effects of GS-3583 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to prematurely discontinue the study, following an internal safety assessment of the molecule, GS-3583.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-496-5657
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — zimberelimab; Cisplatin; Carboplatin; Fluorouracil; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1: Cohort 1: GS-3583 675 μg (Experimental): Participants with advanced solid tumors will receive GS-3583 675 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
  Interventions: Drug: GS-3583
- Part 1: Cohort 2: GS-3583 2000 μg (Experimental): Participants with advanced solid tumors will receive GS-3583 2000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
  Interventions: Drug: GS-3583
- Part 1: Cohort 3: GS-3583 6000 μg (Experimental): Participants with advanced solid tumors will receive GS-3583 6000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
  Interventions: Drug: GS-3583
- Part 1: Cohort 4: GS-3583 12000 μg (Experimental): Participants with advanced solid tumors will receive GS-3583 12000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
  Interventions: Drug: GS-3583
- Part 1: Cohort 5: GS-3583 20000 μg (Experimental): Participants with advanced solid tumors will receive GS-3583 20000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
  Interventions: Drug: GS-3583
- Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy (Experimental): Participants with head and neck squamous cell carcinoma (HNSCC) will receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 21-day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-5-flourouracil (5-FU) 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles.
  Interventions: Drug: GS-3583; Drug: Zimberelimab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy (Experimental): Participants with non-small cell lung cancer (NSCLC) will receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met.
  Interventions: Drug: GS-3583; Drug: Docetaxel
- Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy (Experimental): Participants with HNSCC will receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 21-day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 21-day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles.
  Interventions: Drug: GS-3583; Drug: Zimberelimab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy (Experimental): Participants with HNSCC will receive ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 21-day cycle up to 6 cycles + carboplatin area under th e curve 5 mg/mL/min on Day 1 of each 21-day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles.
  Interventions: Drug: Zimberelimab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy (Experimental): Participants with NSCLC will receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met.
  Interventions: Drug: GS-3583; Drug: Docetaxel
- Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy (Experimental): Participants with NSCLC will receive docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: GS-3583 — Administered as an intravenous (IV) infusion
  Arms: Part 1: Cohort 1: GS-3583 675 μg; Part 1: Cohort 2: GS-3583 2000 μg; Part 1: Cohort 3: GS-3583 6000 μg; Part 1: Cohort 4: GS-3583 12000 μg; Part 1: Cohort 5: GS-3583 20000 μg; Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy
Drug: Zimberelimab — Administered as an IV infusion
  Arms: Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy
Drug: Cisplatin — Administered as an IV infusion
  Arms: Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy
Drug: Carboplatin — Administered as an IV infusion
  Arms: Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy
Drug: 5-Fluorouracil — Administered as an IV infusion
  Arms: Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy
Drug: Docetaxel — Administered as an IV infusion
  Arms: Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy; Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy; Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy

SUMMARY:
This study is planned to be conducted in 2 parts: Part 1: Dose Escalation and Part 2: Safety Run-In and Randomized Expansion.

The primary objectives of Part 1 are 1) To characterize the safety and tolerability of GS-3583 as monotherapy in participants with advanced solid tumors. 2) To determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of GS-3583 as monotherapy in participants with advanced solid tumors.

The primary objectives of Part 2 is to assess the safety and tolerability and to determine the RP2D of GS-3583 in combination with zimberelimab (ZIM) and platinum (cisplatin or carboplatin) + 5-fluorouracil (5-FU) chemotherapy in participants with head and neck squamous cell carcinoma (HNSCC) (Cohort A) or in combination with docetaxel in participants with non-small cell lung cancer (NSCLC) (Cohort B).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumor that is refractory to or intolerant of standard therapy or for which no standard therapy is available
* Have measurable disease on imaging based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
* Eastern Cooperative oncology Group (ECOG) performance status of ≤ 2
* Life expectancy of ≥ 3 months, in the opinion of the investigator
* Adequate organ function as assessed by hematological, renal, and hepatic parameters, and no clinically significant coagulopathy

Key Exclusion Criteria:

* Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery within 3 weeks of Cycle 1 Day 1; a 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with sponsor approval
* Known severe hypersensitivity reactions (NCI CTCAE Grade ≥ 3) to fully human monoclonal antibodies or fusion proteins, GS-3583 formulation excipients, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with corticosteroids, any history of anaphylaxis, or uncontrolled asthma
* Concurrent active malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer who has undergone potentially curative therapy with no evidence of disease. Individuals with other previous malignancies are eligible if disease free for > 2 years.
* Previous history of hematological malignancy, monoclonal gammopathy of unknown significance (MGUS) or other preleukemic states (Presence of clonal hematopoiesis of indeterminate potential (CHIP)/age related clonal hematopoiesis (ARCH) is acceptable)
* Known CNS metastasis(es), unless metastases are treated and stable and the individual does not require systemic corticosteroids for management of CNS symptoms at least 1 week prior to study treatment. Individuals with history of carcinomatous meningitis are excluded regardless of clinical stability.
* Active or history of autoimmune disease that has required systemic treatment within 2 years of the start of study treatment (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)

  * Note: Individuals with diabetes type 1, vitiligo, psoriasis, hypothyroid disease, or hyperthyroid disease, not requiring immunosuppressive treatment are eligible.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - START Midwest, Grand Rapids, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - NEXT oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brody J, Thompson JA, Tolcher AW, Kuhne MR, Huang XR, et al. Phase 1b Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of GS3583, a FLT3 Agonist Fc Fusion Protein, in Patients With Advanced Solid Tumors [Poster TPS3147]. J Clin oncol 2021 June; 39 (15_suppl).
- [Result] Tolcher AW, Brody J, Rajakumaraswamy N, Lakhani NJ, Kuhne MR, Trowe T, et al. Phase 1b study of GS-3583, a novel FLT3 agonist Fc fusion protein, in patients with advanced solid tumors. [Poster TPS2566]. J Clin oncol 2022 June; 40 (16_suppl).
- [Result] Dauki AM, Jones A, Singh I, Rajakumaraswamy N, Qin A, et al. Population pharmacokinetics of GS-3583 in healthy volunteers and patients with advanced solid tumors [Poster II-083]. Clin Pharmacol Ther 2023 March; 113 (S5-S100).
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-496-5657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. This study was planned to be conducted in 2 parts: Part 1: Dose Escalation Part and Part 2: Safety Run-In and Randomized Expansion Part. Due to early termination of the study, Part 2 was not conducted. Results are reported only for Part 1 of the study.
Pre-assignment Details: 22 participants were screened.
Groups:
- Part 1: Cohort 1: GS-3583 675 μg: Prior to the start of enrollment in this study, the GS-3583 dose of 675 µg was evaluated in healthy volunteers in another study, GS-US-496-5619 and deemed well tolerated, therefore, no participants were enrolled at the planned Cohort 1 dose of 675 µg in this study and this cohort was excluded from the study. The enrolment in the study started in Cohort 2 at a dose of 2000 µg.
- Part 1: Cohort 2: GS-3583 2000 μg: Participants received GS-3583 2000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
- Part 1: Cohort 3: GS-3583 6000 μg: Participants received GS-3583 6000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
- Part 1: Cohort 4: GS-3583 12000 μg: Participants received GS-3583 12000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
- Part 1: Cohort 5: GS-3583 20000 μg: Participants received GS-3583 20000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant met study treatment discontinuation criteria.
- Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy: Safety Run-In Cohort A of Part 2 were to include participants with head and neck squamous cell carcinoma (HNSCC) to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + zimberelimab (ZIM) 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of body surface area (BSA) on Day 1 of each 21-day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-flourouracil (5-FU) 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy: Safety Run-In Cohort B of Part 2 were to include participants with non-small cell lung cancer (NSCLC) to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy: Safety Run-In Cohort A of Part 2 were to include participants with HNSCC to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 28- day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy: Randomized Expansion Cohort A of Part 2 were to include participants with HNSCC to receive ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 21-day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 21- day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy: Randomized Expansion Cohort B of Part 2 were to include participants with NSCLC to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy: Randomized Expansion Cohort B of Part 2 were to include participants with NSCLC to receive docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
Period: Overall Study
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Started | 0 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Part 1: Cohort 2: GS-3583 2000 μg: Participants received GS-3583 2000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant meets study treatment discontinuation criteria.
- Part 1: Cohort 3: GS-3583 6000 μg: Participants received GS-3583 6000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant meets study treatment discontinuation criteria.
- Part 1: Cohort 4: GS-3583 12000 μg: Participants received GS-3583 12000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant meets study treatment discontinuation criteria.
- Part 1: Cohort 5: GS-3583 20000 μg: Participants received GS-3583 20000 μg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle for up to 13 cycles (up to 52 weeks) or until the participant meets study treatment discontinuation criteria.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 2 | 1 | 4
  >=65 years | 3 | 2 | 1 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (1.2) | 63 (17.6) | 58 (15.3) | 70 (7.5) | 66 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 1 | 6
  Male | 1 | 0 | 3 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 3 | 1 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any toxicity (hematologic, non-hematologic, dosing/procedures-related toxicities, or grade 5 event (ie death)) occurring with GS-3583 monotherapy during the DLT assessment period (from Day 1 up to Day 28) considered at least possibly related to GS-3583 monotherapy.
Time Frame: Part 1: Day 1 through Day 28; Part 2: Day 1 through Day 21
Population: DLT Evaluable Analysis Set included all participants who were enrolled for dose escalation, received all prescribed treatments and completed safety procedures through DLT assessment period (from Day 1 through Day 28 inclusive of the last day) or experienced a DLT prior to end of DLT assessment period as specified in protocol. No participants were enrolled in Part 2, so, data are reported for Part 1 only.
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy: Safety Run-In Cohort A of Part 2 were to include participants with HNSCC to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 28- day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy: Safety Run-In Cohort B of Part 2 were to include participants with NSCLC to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + docetaxel 75 mg/m^2 on Day 1 of each 21-day cycle until 1 or more criteria for discontinuation are met. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy: Randomized Expansion Cohort A of Part 2 were to include participants with HNSCC to receive GS-3583 at a dose determined in Part 1 on Day 1 of every 21-day cycles for up to 8 cycles + ZIM (ZIm) 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 28- day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
- Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy: Randomized Expansion Cohort A of Part 2 were to include participants with HNSCC to receive ZIM 360 mg, on Day 1 of each 21-day cycle up to 105 weeks + cisplatin 100 mg/m^2 of BSA on Day 1 of each 28- day cycle up to 6 cycles + carboplatin area under the curve 5 mg/mL/min on Day 1 of each 28- day cycle up to 6 cycles + 5-FU 1000 mg/m^2 of BSA/day on Days 1 to 4 of 21-day cycle up to 6 cycles. However, as the study was early terminated, no participants were enrolled in Part 2 of the study.
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants |  | 0 | 0 | 0 | 0 |  |  |  |  |  |

2. Primary Outcome: Parts 1 and 2: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: TEAEs were AEs with onset dates on or after the first dose and up to 90 days after the date of the last dose of study treatment or the day before initiation of subsequent therapy, whichever occurred first. TEAEs severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal. Participants were counted at the highest AE grade experienced.
Time Frame: First dose date up to last dose date plus 90 days (Up to 4 months)
Population: The Safety Analysis Set included all the participants who received at least 1 dose of study drug. No participants were enrolled in Part 2, so, data are reported for Part 1 only.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants |  | 100 | 100 | 100 | 100 |  |  |  |  |  |

3. Primary Outcome: Parts 1 and 2: Percentage of Participants With Laboratory Abnormalities According to the NCI CTCAE Version 5.0
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time, up to 90 days after the last dose of study drug or the day before initiation of subsequent therapy, whichever occurred first. A treatment-emergent laboratory abnormality severity was graded according to the NCI CTCAE version 5.0. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal. Participants were counted at the highest AE grade experienced.
Time Frame: First dose date up to last dose date plus 90 days (Up to 4 months)
Population: The Safety Analysis Set will include all participants who received at least 1 dose of study drug. No participants were enrolled in Part 2, so, data are reported for Part 1 only.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants |  | 100 | 100 | 100 | 100 |  |  |  |  |  |

4. Primary Outcome: Parts 1 and 2: Percentage of Participants With GS-3583 Anti-drug Antibodies (ADAs) at Any Visit
Description: Participants were monitored for the development of ADAs throughout their treatment period with GS-3583 and at the end of study.
Time Frame: Cycles 1and 3,pre-dose,End of Infusion (EOI);2,6 hours;Days 2,3,5,8,15 post Day 1EOI;Day 15:Cycle 1:predose and EOI;2 hours post EOI;Cycle 3:336 hours and Day 24 post EOI(Cycle length = 28 days in Part 1; 21 days for Part 2;infusion duration=60 minutes)
Population: Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of study drug and have at least 1 non-missing ADA test result. No participants were enrolled in Part 2, so, data are reported for Part 1 only.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants |  | 33.3 | 33.3 | 0 | 0 |  |  |  |  |  |

5. Secondary Outcome: Part 1: Pharmacokinetic (PK) Parameter: AUCtau of GS-3583
Description: AUCtau is defined as the area under the concentration versus time curve over the dosing interval where tau = 15 days.
Time Frame: Cycles 1 and 3, pre-dose, EOI; 2, 6 hours; Days 2, 3, 5, 8, 15 post Day 1 EOI; Day 15:Cycle 1:predose and EOI; 2 hours post EOI;Cycle 3:336 hours and Day 24 post EOI (Cycle length for all cycles=28 days in Part 1; Infusion duration=60 minutes)
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of study drug and have at least 1 non-missing postdose concentration value reported by the PK laboratory. Data for Cycle 3 is not reported due to participant's confidentiality reasons, as there was only 1 or 2 participants in each of these groups during Cycle 3.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4
h*ng/mL
  Cycle 1 |  | 82100 (19900) | 249000 (124000) | 352000 (41300) | 832000 (223000)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part 1: PK Parameter: Cmax of GS-3583
Description: Cmax is defined as the maximum observed plasma concentration.
Time Frame: Cycles 1 and 3,pre-dose,EOI;2, 6 hours;Days 2, 3, 5, 8, 15 post Day 1 EOI;Day 15:Cycle 1:predose and EOI;2 hours post EOI;Cycle 3:336 hours and Day 24 post EOI (Cycle length for all cycles=28 days in Part 1;Infusion duration=60 minutes)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4
ng/mL
  Cycle 1 |  | 643 (36.3) | 1860 (562) | 2520 (244) | 5800 (1460)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Part 1: PK Parameter: Tmax of GS-3583
Description: Tmax is defined as the time to reach maximum observed plasma concentration (Tmax).
Time Frame: Cycles 1 and 3, pre-dose, EOI; 2, 6 hours; Days 2, 3, 5, 8, 15 post Day 1 EOI; Day 15:Cycle 1:predose and EOI; 2 hours post EOI; Cycle 3:336 hours and Day 24 post EOI (Cycle length for all cycles=28 days in Part 1; infusion duration=60 minutes)
Population: as for outcome 5
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 4
hours (h)
  Cycle 1 |  | 1.1 [1.0 to 1.1] | 2.0 [1.1 to 5.6] | 1.1 [1.1 to 2.0] | 1.7 [1.2 to 2.1]
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Part 2: Confirmed Objective Response Rate (ORR)
Description: Confirmed ORR is defined as the percentage of participants who have achieved confirmed CR or PR according to RECIST V1.1 and assessed by the investigator. Per RECIST V1.1, CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: First dose date in Part 2 to End of Study (approximately 4.2 months)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose date until first date of disease progression (PD) or death from any cause, whichever comes first as measured per RECIST V1.1 as assessed by the investigator. Per RECIST V1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: First dose date in Part 2 to End of Study (approximately 4.2 months)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: DOR was defined as time of first response (CR or PR) per RECIST V1.1 as assessed by the investigator until the date of first documented disease progression or death, whichever comes first. Per RECIST V1.1, CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: First dose date in Part 2 to End of Study (approximately 4.2 months)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 2: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death from any cause.
Time Frame: First dose date in Part 2 to End of Study (approximately 4.2 months)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part 2: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with a best overall confirmed response of CR or PR or stable disease. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: First dose date in Part 2 to End of Study (approximately 4.2 months)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part 2: PK Parameters: Cmax for GS-3583
Description: Cmax is defined as the maximum observed serum concentration of drug.
Time Frame: Safety-run In:Cycles 1 and 3: Day 1, predose, EOI; 2, 6 hours, Days 8, 15; Part 2 all arms:Cycles 2 and 5: Day 1 predose, EOI and every odd cycles; 60-day FU; (Cycle length of all cycles = 21 days in Part 2; Infusion duration=60 minutes)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Part 2: PK Parameter: Tmax for GS-3583
Description: Tmax is defined as the time (observed time point) of the occurrence of Cmax.
Time Frame: Safety-run In: Cycles 1, and 3: Day 1, predose, EOI; 2, 6 hours, Days 8, Day 15; Part 2: all arms: Cycles 2 and 5: Day 1 predose, EOI and every odd cycles; 6-day FU; (Cycle length of all cycles = 21 days in Part 2; Infusion duration=60 minutes)
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Part 2: PK Parameter: AUCtau of GS-3583
Description: AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
Time Frame: as for outcome 14
Population: No participants were enrolled in Part 2 of the study, so, data was not collected for this outcome measure.
Arm/Group | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14.8 months
Description: All-Cause Mortality: All Enrolled Analysis Set included all participants who received a study participant identification number in the study after screening.
  Adverse Events: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Part 1: Cohort 1: GS-3583 675 μg | Part 1: Cohort 2: GS-3583 2000 μg | Part 1: Cohort 3: GS-3583 6000 μg | Part 1: Cohort 4: GS-3583 12000 μg | Part 1: Cohort 5: GS-3583 20000 μg | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 3/3 | 2/3 | 2/3 | 2/4 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/3 | 1/3 | 2/3 | 1/4 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 3/3 | 3/3 | 4/4 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: GS-3583 675 μg (N=0) | Part 1: Cohort 2: GS-3583 2000 μg (N=3) | Part 1: Cohort 3: GS-3583 6000 μg (N=3) | Part 1: Cohort 4: GS-3583 12000 μg (N=3) | Part 1: Cohort 5: GS-3583 20000 μg (N=4) | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy (N=0)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: GS-3583 675 μg (N=0) | Part 1: Cohort 2: GS-3583 2000 μg (N=3) | Part 1: Cohort 3: GS-3583 6000 μg (N=3) | Part 1: Cohort 4: GS-3583 12000 μg (N=3) | Part 1: Cohort 5: GS-3583 20000 μg (N=4) | Part 2: Safety Run-In Cohort A: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Safety Run-In Cohort B: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort A: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort A: Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort B: GS-3583 + Combination Anticancer Therapy (N=0) | Part 2: Randomized Expansion Cohort B: Combination Anticancer Therapy (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT04747470/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04747470/SAP_001.pdf